CLINICAL TRIAL: NCT01595646
Title: Study of Nasal Insulin to Fight Forgetfulness - Long-acting Insulin Detemir - 120 Days (SL120)
Acronym: SL120
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00023230; ZEN-10-173646US (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2018-04

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Memory; Intranasal insulin; Alzheimer's disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Sodium Chloride; Saline Solution; Insulin Detemir; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saline (Placebo Comparator): Saline placebo taken twice per day via intranasal route.
  Interventions: Drug: Saline
- Insulin Detemir (Experimental): 20IU of Insulin Detemir taken twice per day (40IU total per day) via intranasal route
  Interventions: Drug: Insulin detemir
- Insulin (Experimental): 20IU Insulin, administered twice per day (40IU total per day) via intranasal route
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Saline — Saline, administered intranasally twice per day for a 16 week duration
  Other Names: Saline solution
  Arms: Saline
Drug: Insulin detemir — 20IU of insulin detemir, administered intranasally twice per day for a 16 week duration (total of 40IU insulin detemir per day)
  Other Names: Levemir
  Arms: Insulin Detemir
Drug: Insulin — 20IU insulin, administered intranasally twice per day for a 16 week duration (total of 40IU insulin per day)
  Other Names: Novolin R
  Arms: Insulin

SUMMARY:
The study will examine the effects of intranasally administered long-acting insulin detemir on cognition in persons with Alzheimer's disease (AD) or amnestic mild cognitive impairment (aMCI). The rationale for these studies is derived from growing evidence that insulin contributes to multiple brain functions, and that insulin dysregulation can contribute to AD pathogenesis. Thus, therapies aimed at restoring normal insulin signaling in the CNS may have beneficial effects on brain function. Intranasal administration of insulin increases insulin signaling in the brain without raising peripheral levels and causing hypoglycemia. Insulin detemir is an insulin analogue that may have better action in brain than other insulin formulations because of its albumin binding properties. The investigators will test the therapeutic effects of intranasally-administered insulin detemir in a study in which participants will receive insulin detemir, regular insulin, or placebo over a four month period. The investigators will test the hypothesis that insulin and insulin detemir will both improve memory and daily functioning in persons with AD/aMCI compared with placebo, but that insulin detemir will have the greatest effect.

DETAILED DESCRIPTION:
It is well-known that insulin, a hormone that is naturally secreted by the pancreas, plays an important physiological role by regulating blood sugar levels in the body. Researchers now know that insulin plays many important roles in the brain as well. Insulin seems to be especially active in the part of the brain that corresponds to learning and memory. Studies have shown that when people have insufficient insulin in the brain (which, for example, is the case with Type-II diabetes), they are increasingly at risk to develop memory problems and Alzheimer's disease. In a past study, the investigators administered intravenous insulin to participants and found that it improves memory. However, that particular method would not be a practical intervention for people with Alzheimer's disease due to the risks of hypoglycemia or exacerbation of insulin resistance. Instead, the investigators use an "intranasal" method of administration, in which the insulin is inserted into a device, and administered intranasally. In this method, the insulin travels directly to the brain, and bypasses the body. Past studies have also demonstrated that this can be a reliable way to improve memory, and it does not change the body's blood glucose levels.

In our past studies, investigators have used regular insulin, which lasts about 3-4 hours and creates a similar "spike" in insulin that one would have after eating a meal. However, in normal physiology, the pancreas also releases small and more constant "pulses" of insulin throughout the day and night, establishing a base level of insulin. Accordingly, several longer-lasting types of insulin are now available that last closer to 10-12 hours, mimicking that basal level of insulin. The current study uses a long-lasting type of insulin called "insulin detemir," to determine if learning and memory will benefit from a more consistent supplement of insulin. The investigators want to determine whether this treatment can benefit people who already have a memory impairment-either they have a diagnosis of Alzheimer's disease (AD) or have a mild cognitive impairment (MCI), a condition that precedes Alzheimer's disease. The investigators will examine cognition, daily function, cerebral blood flow, and different markers of Alzheimer's disease that are in the blood and cerebral spinal fluid (CSF) as outcome measures.

The investigators have these specific aims:

1. We will test the hypothesis that compared to placebo, four months of treatment with intranasal insulin or insulin detemir will improve cognition and function in adults with AD or MCI, but that greater effects will be observed for insulin detemir.
2. We will examine the effects of intranasal insulin and insulin detemir on cerebral blood flow in adults with AD or MCI.
3. We will examine the effects of intranasal insulin and insulin detemir on CSF Aβ, tau and inflammatory markers in adults with AD or MCI.

To examine these hypotheses, the investigators are recruiting approximately 90 participants who have been diagnosed with AD or mild cognitive impairment. They will be randomly selected to take a placebo (saline), insulin detemir, or insulin. Cognition, the level of daily functioning, glucose tolerance, and cerebral blood flow will be tested before they begin the study drug, and after 16 weeks of the study drug. Some participants will also undergo a lumbar puncture both before beginning study drug and after 16 weeks of taking the study drug.

Statistical analysis will follow an intent-to-treat (ITT) approach; that is, subjects will be analyzed in their original randomized group regardless of adherence to group assignment. A completer analysis will also be performed, including only those subjects who successfully complete the treatment phase. Missing data will be handled using multiple imputation linear regression. We will conduct secondary analyses on other measures of cognition, daily function, cerebral blood flow, and CSF biomarkers. For ASL-MRI, following coregistration and processing, parametric maps will be generated to determine regional CBF values by treatment group. Secondary analyses will also examine treatment duration (2-month vs. 4-month) for all relevant outcomes. All models will be adjusted for age and an index of peripheral insulin sensitivity (derived from 120-minute OGTT glucose and insulin values) if statistically warranted, and posthoc contrasts will be performed when appropriate. Secondary analyses will also evaluate whether treatment response of cognition, daily function, CSF and plasma markers, and insulin differ according to APOE4 genotype. Although these analyses will be exploratory due to possible limited APOE4 by treatment arm cell size, the data will be examined for statistical trends that warrant further exploration in larger trials. Other secondary analyses will examine associations among treatment-related outcomes using scores derived from multiple regression of data collected during the treatment phase residualized with respect to baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-89
* Diagnosed with mild cognitive impairment, or mild/moderate AD

Exclusion Criteria:

* Excessively high or low blood pressure, heart rate
* Pre-existing diabetes not controlled by exercise/diet
* Previous/current use of insulin
* Significant elevations in lipids, liver enzymes
* Menstrual period within the last 12 months
* Significant neurological or medical disorder (other than AD)
* Significant use of nasal decongestants
* Current use of anti-psychotic, anti-convulsive, anxiolytic, glucocorticoids, or sedative medications

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-03-12 (Actual); Study Completion 2015-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - VA Puget Sound Health Care System - American Lake Division, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Detemir: 20IU of Insulin Detemir taken twice per day (40IU total per day)
  Insulin detemir: 20IU of insulin detemir, administered intranasally twice per day for a 16 week duration (total of 40IU insulin detemir per day)
- Insulin: 20IU Insulin, administered twice per day (40IU total per day)
  Insulin: 20IU insulin, administered intranasally twice per day for a 16 week duration (total of 40IU insulin per day)
Period: Overall Study
Arm/Group | Saline | Insulin Detemir | Insulin
Started | 13 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Insulin Detemir | Insulin | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 3 | 11
  >=65 years | 8 | 8 | 9 | 25
Age, Continuous [Mean (Full Range); unit: years] | 68 [61 to 75] | 66 [62 to 70] | 68 [56 to 80] | 68 [56 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 7 | 19
  Male | 6 | 6 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 12 | 12 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Verbal Memory Composite
Description: The composite will consist of the sum of Z scores for Delayed Story Recall and Buschke Selective Reminding Test. In the Story Recall test subjects listen to a story containing 44 informational bits that is read once. Subjects will be asked to recall the story immediately after the reading and after a 20-min delay. Credit is awarded for each bit recalled verbatim or accurately paraphrased. The Buschke Selective Reminding Test measures verbal memory through multiple trials of a list learning task. A list of 12 words is audibly presented to the subject, and subjects recall as many words as possible. On subsequent trials, subjects are only told those words they omitted on the previous trial. The procedure continues until the subject recalls all words on two successive trials or to the twelfth trial. After a 30-minute delay, subjects recall as many items as possible. Number of items recalled after the delay will be summed. Higher scores indicate better performance.
Time Frame: Change from Baseline in Verbal Memory at 16 weeks
Population: The study is in data analysis and manuscript write-up.
Measure: Mean (Standard Error); unit: Change in Z score memory composite
Arm/Group | Saline | Insulin Detemir | Insulin
Number analyzed (Participants) | 12 | 12 | 12
Change in Z score memory composite | -.31247583 (.23) | .33390008 (.23) | -.05181561 (.22)

2. Secondary Outcome: Cerebral Spinal Fluid (CSF) Biomarkers of AD
Description: CSF Abeta (Abeta 42) and Tau (total tau and phosphorylated tau) will be measured in each subject.
Time Frame: Change from Baseline in CSF Biomarkers at 16 Weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Saline | Insulin Detemir | Insulin
Number analyzed (Participants) | 12 | 12 | 12
pg/mL
  Abeta42 Pre | 331.5 (148.4) | 408.5 (196.9) | 305.5 (86.1)
  Abeta 42 Post | 384 (212) | 381.8 (227.8) | 325 (92.1)
  Tau Pre | 109.7 (27) | 118.3 (49.1) | 132.3 (71)
  Tau Post | 117.1 (36.8) | 107.6 (56) | 152.2 (106.7)
  Tau-P181 Pre | 65.1 (33.1) | 63.9 (28) | 74 (28.9)
  Tau-P181 Post | 72.17 (25.3) | 64.1 (19.8) | 68.5 (39.7)

3. Secondary Outcome: Cerebral Spinal Fluid (CSF) Biomarkers of AD TTau-P181/Abeta42 Ratio
Description: CSF Abeta (ABeta 38, ABeta 40, and Abeta 42) and Tau (total tau and phosphorylated tau) will be measured in each subject. A pre and post ratio of TTau-P181/Abeta42 will be given.
Time Frame: Change from Baseline in CSF Biomarkers at 16 Weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Saline | Insulin Detemir | Insulin
Number analyzed (Participants) | 12 | 12 | 12
ratio
  TTau-P181/Abeta42 ratio Pre | .27 (19) | .23 (.22) | .27 (.14)
  Tau-P181/Abeta42 ratio Post | .30 (.21) | .23 (.16) | .23 (.13)

4. Secondary Outcome: Functional Ability
Description: Subjects will have a collateral informant (i.e., spouse or friend) rate the subjects' ability to carry out activities of daily living on the Dementia Severity Rating Scale. The Dementia Severity Rating Scale is made up of sub-scales and the scores from each are summed to produce one score. The scale assess memory, ability to get from place to place, and speech and language each with a range from 0-6; recognition of family members and social and community both having a range from 0-5; orientation of time, orientation to place, ability to make decisions, home activities and responsibilities, and control of urination and bowels each having a range of 0-4; personal care- cleanliness and eating both with a range of 0-3. The total score range is from 0-54 and lower scores denotes better outcomes.
Time Frame: baseline, month 2, and month 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Insulin Detemir | Insulin
Number analyzed (Participants) | 12 | 12 | 12
units on a scale
  Baseline | 7.3 (6.9) | 8.7 (6.7) | 7.7 (6.8)
  month 2 | 7 (6.7) | 9.7 (7.3) | 9.7 (7.4)
  month 4 | 6.9 (7.1) | 9.1 (7.5) | 10.6 (9.4)

5. Secondary Outcome: The Alzheimer's Disease Assessment Scale-Cognitive [ADAS-Cog/Alzheimer's Disease Cooperative Study (ADCS)] - MCI Revision
Description: This cognitive screening measure contains measures of confrontational naming, following commands, constructional praxis, ideational praxis, orientation, and language production and comprehension. Total scores range from 0-70, with higher scores indicating greater cognitive impairment.
Time Frame: Baseline, Month 2 and Month 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Insulin Detemir | Insulin
Number analyzed (Participants) | 12 | 12 | 12
units on a scale
  Baseline | 20 (11.7) | 21.6 (13.7) | 19.8 (12.8)
  Month 2 | 18.5 (11.8) | 23.4 (17.1) | 21.8 (13.6)
  Month 4 | 20.4 (13.7) | 19.5 (12.9) | 22.6 (15.8)

6. Other Pre Specified Outcome: Executive Function Composite
Description: Sum of Z Scores from Dot Counting Test (test of executive functioning) and Benton Visual Retention Test Form F&G (a test of visual working memory)
Time Frame: Change from Baseline in Executive Functioning at 16 Weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Plasma Biomarkers of AD
Description: Plasma Abeta (ABeta 38, ABeta 40, and Abeta 42) and Tau (total tau and phosphorylated tau) will be measured in each subject.
Time Frame: Change from Baseline in Plasma Biomarkers at 16 Weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Cerebral Blood Flow
Description: Functional MRI and arterial-spin labeling perfusion MRI
Time Frame: Change from Baseline in Cerebral Blood Flow at 16 Weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Glucose Tolerance
Description: Subjects will undergo oral glucose tolerance test (OGTT) to assess glucose tolerance
Time Frame: Change from Baseline in Glucose Tolerance at 16 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Saline | Insulin Detemir | Insulin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 0/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=12) | Insulin Detemir (N=12) | Insulin (N=12)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — PT experienced chest pain during MRI.
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — PT began to feel some anxiety during the MRI scan.
Congestion (General disorders) | 1 (1) | 0 (0) | 0 (0) — PT reported head congestion.
Cold & Flu Symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) — PT reported having symptoms resembling a cold or flu.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No